CLINICAL TRIAL: NCT04964180
Title: Rectal Indomethacin Versus Intraperitoneal Lidocaine for Analgesia After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Gad Sayed Gad, assisstant professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: analgesia LC
Record Dates: First submitted 2021-07-01; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indomethacin group (Active Comparator): group indomethacin (40 patients) recived two 100 mg indomethacin rectal suppositories 2 hours prior to surgery
  Interventions: Drug: Indomethacin suppository
- intraperitoneal lidocaine (Active Comparator): 200 ml saline containing 200 mg 2%lidocaine immediately after abdominal cO2 insufflation( pneumoperitoneum) the surgeon sprayed the total solution on the upper surface of the liver under the right subdiaphragmatic space, left subdiaphragmatic space and around the cholecystectomy site , all patients were maintained in trendelenberg position
  Interventions: Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Indomethacin suppository — two 100 mg indomethacin rectal suppositories 2 hours prior to surgery
  Other Names: Indocid suppository
  Arms: indomethacin group
Drug: Lidocaine 2% Injectable Solution — 200 ml saline containing 200 mg 2%lidocaine intraperitoneal insilltation
  Other Names: lidocaine HCL 2%
  Arms: intraperitoneal lidocaine

SUMMARY:
Hospitals, Qena, Egypt in period between May 2020 to May 2021.eighty patients was scheduled to elective laparoscopic cholecystectomy , divided Into two groups randomly using closed envelop method. Group IP lidocaine(40 patients ) received 200 ml saline containing 200 mg 2%lidocaine immediately after abdominal cO2 insufflation( pneumoperitoneum) the surgeon sprayed the total solution on the upper surface of the liver under the right subdiaphragmatic space, left subdiaphragmatic space and around the cholecystectomy site , all patients were maintained in trendelenberg position.

At the end of the laparoscopic procedure, group indomethacin (40 patients) recived two 100 mg indomethacin rectal suppositories 2 hours prior to surgery

ELIGIBILITY:
Inclusion Criteria:

* .ASA physical status 1-2 patients.
* 18-60 years old .

Exclusion Criteria:

* using or allergic to nonsteroidal anti inflammatory drugs (NSAIDs) or aspirin .
* history of serious hepatic disease.
* renal or gastrointestinal disease.
* bleeding disorder.
* body mass index BMI <18 or ˃30 m2/kg.
* history of abdominal surgery or chronic pain disorder other than gallbladder.
* disease or allergy to lidocaine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
VAS scores postoperative | 24 hours posoperative
  a standard 10-cm VAS was used, where one end of the scale represented no pain (0 cm), and the other end the most severe pain imaginable (10 cm), the distance in centimeters being taken as the pain score
postoperative opoiods analgesics requirements | 24 hours postoperative
  we used (iv pethidine )whenever the patient complained of pain. IV pethidine injection 25-50 mg was given as rescue analgesic whenever the patient experienced pain ≥ to 5 VAS

SECONDARY OUTCOMES:
Pain starting time after surgery and Pethidine required first time. | 24 hours postoperative
  Pain starting time after surgery and Pethidine required first time.

CONTACTS AND LOCATIONS:
Locations (1):
- Gad sayed Gad, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided